CLINICAL TRIAL: NCT01334138
Title: Effect of Dietary Sodium Intake on Blood Pressure in Hypertensive Patients in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/233
Record Dates: First submitted 2011-04-11; First posted 2011-04-12 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Arterial Hypertension
Keywords: hypertension; sodium; diet
MeSH Terms: conditions — Hypertension | interventions — Diet; Sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 4-week diet, low in sodium (Experimental): The study subjects go on a 4-week diet, low in sodium.
  Interventions: Other: A 4-week diet, low in sodium.

INTERVENTIONS:
Other: A 4-week diet, low in sodium. — Study subjects receive personal advice to decrease sodium consumption and will change his diet for 28 days.
  Follow up is performed by measuring blood pressure, a 24-hour urine sample collection, diaries and questionnaires.

SUMMARY:
There is strong evidence that our current consumption of salt is the major factor increasing blood pressure (BP). The current salt intake in most countries in the world is 9 to 12 grams per day (g/d), whil the World Health Organization's recommendation is < 5 g/d.

The aims of the present study is to determine if the overconsumption of salt influences the bp in patients with uncontrolled hypertension or frequently elevated bp.

Each study subject will complete questionnaires, and their usual dietary salt intake is estimated from food composition on 3 completed food diaries. This is also compared with a 24-hour urine sample collection.

Based on these results, the study subject receives personal advice to decrease sodium consumption and will change the diet for at least 28 days. During this diet, bp will be measured and food diaries will be completed. After the intervention, a questionnaire and a 24-hour urine sample collection will be collected.

ELIGIBILITY:
Inclusion Criteria:

* adults, 50 years of age or older with changing blood pressure (bp) with or without drugs and patients with uncontrolled bp despite drugs
* An average systolic bp on 2 of the 3 previous visits of 140 mm Hg or more (130 mm Hg for diabetics) and an average diastolic bp of 80 to 100 mm Hg.
* Blood analysis (fasting glycaemia, creatinin, total cholesterol, high- density lipoprotein cholesterol) in the last 6 months
* At least 3 criteria of the following:

  * using table salt
  * 2-3/weeks consumption of prepared meals (butchery, warehouse...)
  * 2-3/weeks consumption of effervescent tablet
  * Daily consumption of cheese/cold cuts
  * Daily consumption of salted butter/margarine
  * 2-3/weeks consumption of smoked fish/meat
  * 2-3/weeks consumption of bouillon cube-soup (self-made or preserved)
  * 2-3/weeks consumption of cookies
  * 2-3/weeks consumption of vegetables preserved in jars
  * 2-3/weeks consumption of vegetable juice
  * 2-3/weeks consumption of snacks (chips, cheese, nuts...)

Exclusion Criteria:

* heart failure
* renal insufficiency
* secondary hypertension
* isolated systolic/diastolic hypertension
* bp difference of more than 10 mm Hg between left and right arm
* lactation or pregnancy
* active malignancy
* an active 'low in salt' diet
* changing the use of antihypertensive drugs or other medication that would affect bp for the last 4 weeks
* impaired cognitive functioning$
* planning a smoke cessation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Measurement of blood pressure after a 4-week diet, low in sodium. | after 4 weeks

SECONDARY OUTCOMES:
Life style change after a 4-week diet, low in sodium. | after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan Dehenauw, Ph.D, Professor, Principal Investigator — University Ghent
Locations (1):
- University Ghent, Ghent, Belgium